CLINICAL TRIAL: NCT03924284
Title: Evaluation of Novel Molecular Assays for the Detection of Influenza Virus
Brief Title: Novel Assays for Detection of Influenza Virus
Status: Withdrawn | Type: Observational
Why Stopped: Wrong entry
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Kelvin Kai-Wang To, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: FluA_20190110
Record Dates: First submitted 2019-01-11; First posted 2019-04-23 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Influenza A Virus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The total nucleic acid will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NPA positive: NPA specimens that are tested positive for influenza A virus by commercially available assay or by the Public Health Laboratory Services Branch of Hong Kong
  Interventions: Diagnostic Test: PB2 gene RT-PCR; NS gene RT-PCR
- NPA negative: NPA specimens that are tested negative for influenza A virus by commercially available assay or by the Public Health Laboratory Services Branch of Hong Kong
  Interventions: Diagnostic Test: PB2 gene RT-PCR; NS gene RT-PCR
- Saliva positive: Saliva specimens that are tested positive for influenza A virus by commercially available assay or by the Public Health Laboratory Services Branch of Hong Kong
  Interventions: Diagnostic Test: PB2 gene RT-PCR; NS gene RT-PCR
- Saliva negative: Saliva specimens that are tested negative for influenza A virus by commercially available assay or by the Public Health Laboratory Services Branch of Hong Kong
  Interventions: Diagnostic Test: PB2 gene RT-PCR; NS gene RT-PCR

INTERVENTIONS:
Diagnostic Test: PB2 gene RT-PCR; NS gene RT-PCR — PB2 gene RT-PCR: RT-PCR targeting the PB2 gene of influenza A virus NS gene RT-PCR: RT-PCR targeting NS gene of influenza A virus

SUMMARY:
Seasonal influenza virus causes an estimated 0.3-0.6 million deaths per year. Avian influenza virus H5N1, H7N9 and H5N6 has fatality rate of over 30%. Swine influenza viruses from pigs have also infected humans.

Molecular assays are now used routinely in the detection of influenza viruses. The M gene is often used as the target for all influenza A viruses because the nucleotide sequence of this gene is relatively conserved among all the influenza A viruses. The World Health Organization and the US Centers for Disease Control and Prevention (CDC) have published protocols for molecular detection of influenza A virus M gene.

However, recent studies have shown that mutations in the M gene have led to a reduced sensitivity of RT-PCR assay targeting this gene. Therefore, it is important to use alternative conserved genes as the target of RT-PCR. In this study, our aim is to evaluate two new RT-PCR assays that are based on PB2 and NS gene segment.

DETAILED DESCRIPTION:
I. Background

* Seasonal influenza virus causes an estimated 0.3-0.6 million deaths per year. Avian influenza virus H5N1, H7N9 and H5N6 has fatality rate of over 30%. Swine influenza viruses from pigs have also infected humans.
* Molecular assays are now used routinely in the detection of influenza viruses. The M gene is often used as the target for all influenza A viruses because the nucleotide sequence of this gene is relatively conserved among all the influenza A viruses. The World Health Organization and the US Centers for Disease Control and Prevention (CDC) have published protocols for molecular detection of influenza A virus M gene.
* However, recent studies have shown that mutations in the M gene have led to a reduced sensitivity of RT-PCR assay targeting this gene. Therefore, it is important to use alternative conserved genes as the target of RT-PCR. In this study, our aim is to evaluate two new RT-PCR assays that are based on PB2 and NS gene segment

II. Study objective -To evaluate the sensitivity and specificity of 2 new RT-PCR assays

III. Overall study design

* The investigators will randomly retrieve archived nasopharyngeal and saliva specimens that were previously tested for influenza A virus using commercially available assays in our laboratory, tested for influenza A virus at the Public Health Laboratory Service Branch in Hong Kong. These specimens will be tested for influenza A virus by 4 different RT-PCR assays as listed below:

  1. Our new RT-PCR assay targeting PB2 gene
  2. Our new RT-PCR assay targeting NS gene
  3. M gene RT-PCR published by the World Health Organization
  4. M gene RT-PCR published by the US CDC

     Sensitivity, specificity, positive predictive value and negative predictive value will be determined.

     IV. Nucleic acid extraction and real-time reverse transcription-polymerase chain reaction (RT-PCR) for influenza A virus
* Saliva and nasopharyngeal specimens will be subjected to total nucleic acid (TNA) extraction by NucliSENS easyMAG (BioMerieux, Boxtel, Netherlands).
* Monoplex real-time RT-PCR assays for influenza A virus will be performed. The primers and probes for the M gene RT-PCR have been published by the WHO and the US CDC.

V. Sample size:

* The investigators will perform all 4 RT-PCR assays on a total of 320 specimens, including
* 80 nasopharyngeal specimens which tested positive for influenza A by commercially-available molecular assays or by testing performed at the Public Health Laboratory Services Branch in Hong Kong
* 80 nasopharyngeal specimens which tested negative for influenza A by commercially-available molecular assays or by testing performed at the Public Health Laboratory Services Branch in Hong Kong
* 80 saliva specimens which tested positive for influenza A by commercially-available molecular assays
* 80 saliva specimens which tested negative for influenza A by commercially-available molecular assays

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal or saliva specimens of patients in Queen Mary Hospital of Hong Kong
* Tested for influenza A virus using a commercially available assay or by the Public Health Laboratory Services Branch in Hong Kong

Exclusion Criteria:

* Insufficient specimen volume

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These archived nasopharyngeal and saliva specimens are collected from patients in Queen Mary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-18 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
RT-PCR result | Through study completion, an average of 2 months
  The result of RT-PCR can be positive or negative

SECONDARY OUTCOMES:
Cycle threshold value | Through study completion, an average of 2 months
  The cycle threshold is a surrogate for viral load

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin To, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03924284/Prot_000.pdf